CLINICAL TRIAL: NCT07326644
Title: Effect of Gestational Weight Gain on Regional Anesthesia in Cesarean Patients
Brief Title: Effect of Gestational Weight Gain on Spinal Anesthesia in Elective Cesarean Delivery
Acronym: GWG-CESA
Status: Recruiting | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Sait Fatih Öner, MD, PhD, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: FSH-NEC-GWG-CS-2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gestational Weight Gain; Regional Anesthesia; Cesarean Delivery
Keywords: Gestational weight gain; Spinal anesthesia; Cesarean delivery; Hemodynamic response
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inadequate Gestational Weight Gain: Pregnant women whose gestational weight gain is below the recommended range according to the Institute of Medicine (IOM) 2009 guidelines.
- Adequate or Excessive Gestational Weight Gain: Pregnant women whose gestational weight gain is within or above the recommended range according to the Institute of Medicine (IOM) 2009 guidelines.

SUMMARY:
This prospective, observational, non-interventional study aims to evaluate the effect of gestational weight gain on regional anesthesia characteristics in pregnant women undergoing elective cesarean delivery. No additional intervention, medication, or procedure beyond routine clinical care will be performed. Participants will be classified according to gestational weight gain categories based on the Institute of Medicine (IOM) 2009 guidelines, and spinal anesthesia block characteristics, hemodynamic responses, and perioperative outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-45 years

  * Single pregnancy
  * Planned elective cesarean section
  * Spinal anesthesia (regional anesthesia technique)
  * Pre-pregnancy weight information available (maternal health record, e-Nabız or file record)
  * Recorded pre-delivery weight information
  * Gestational weight gain (GWG) calculable according to the IOM 2009 classification
  * ASA I-II pregnant women
  * Voluntary participation in the study and informed consent

Exclusion Criteria:

* Pregnant women with preeclampsia, severe preeclampsia, eclampsia, or HELLP syndrome

  * Pregnant women with a history of gestational diabetes or pregestational diabetes
  * Multiple pregnancy (twins, triplets, etc.)
  * Preterm pregnancy (<37 weeks)
  * Failure of spinal anesthesia or need for conversion to general anesthesia
  * Lack of pre-pregnancy weight information or weight gain data during pregnancy
  * Pregnancies with fetal anomalies
  * Morbid obesity (BMI ≥ 45 kg/m²)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of pregnant women aged 18 to 45 years who are scheduled for elective cesarean delivery under regional (spinal) anesthesia. All participants will be followed prospectively, and no additional intervention beyond routine clinical care will be performed. Gestational weight gain will be calculated using pre-pregnancy and pre-delivery weight records and classified according to the Institute of Medicine (IOM) 2009 guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-03-05 (Estimated); Study Completion 2026-03-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Spinal Anesthesia-Induced Hypotension | During cesarean delivery (first 20 minutes after spinal anesthesia)
  Occurrence of hypotension following spinal anesthesia, defined as a decrease in mean arterial pressure of ≥20% from baseline or an absolute mean arterial pressure <65 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- Fethi Sekin City Hospital, Elâzığ, Elaziğ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No